CLINICAL TRIAL: NCT06269029
Title: Effect of Chest Mobility Exercises Versus Proprioceptive Neuromuscular Facilitation in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Chest Mobility Exercises Versus Proprioceptive Neuromuscular Facilitation in Patients With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Isaac Zakaria Zarii Yanii, Doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.Rec/012/004297
Record Dates: First submitted 2024-01-17; First posted 2024-02-21 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Chronic Obstructive Pulmonary Disease Moderate
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with COPD assigned for chest mobility (Experimental): This study will be carried on 30 patients with Chronic obstructivepulmonarydisease. Patients will be selected from department (3) Kaser EL-Ainy, Cairo University.
  Interventions: Other: Chest mobility exercises
- patients with COPD assigned for PNF (Experimental): This study will be carried on 30 patients with Chronicobstructivepulmonarydisease. Patients will be selected from department (3) Kaser EL-Ainy, Cairo University.
  Interventions: Other: proprioceptive neuromuscular facilitation

INTERVENTIONS:
Other: Chest mobility exercises — exercises were repeated 6 times on each side with rest of period for 30 seconds in between. The intervention will be carried out for one week with total of 7 sessions. Each Exercise will be accompanied by breathing pattern. In neutral position of exercises, subjects will be asked to exhale during flexion, turning or extension subject will be asked to do inhale.
  Arms: patients with COPD assigned for chest mobility
Other: proprioceptive neuromuscular facilitation — The technique used in this study Proprioceptive neuromuscular facilitation technique of hold and relax stretching for isolated clavicular head of the pectoralis major muscle. The subjects sitting on a chair with back support to keep spine in a neutral position and both their arms are extended and hands are placed behind the occipital region. His both arms will be positioned in glenohumeral horizontal extension, and glenohumeral abduction and external rotation with elbow bent to perform stretch position of pectoral muscle. Then ask him to contract the pectoral muscles .This isometric contraction is held for 6 seconds. The patient then relaxed and passive stretch in the opposite direction . and it was repeated 6 times with rest period 30 seconds. The session will be given every day for one week
  Arms: patients with COPD assigned for PNF

SUMMARY:
Chest mobility exercise versus proprioceptive neuromuscular facilitation in patients with chronic obstructive pulmonary disease

DETAILED DESCRIPTION:
The purpose of this study is designed to compare the therapeutic effect of chest mobility exercises and proprioceptive neuromuscular facilitation stretching on improving chest expansion and functional capacity in patients with chronicobstructivepulmonarydisease?

ELIGIBILITY:
Inclusion Criteria:

All patients will have the following criteria:

1. Age: 50-60 years old
2. All patients will be in mild to moderate of COPD. In accordance with criteria of Global Initiative for Chronic Obstructive Lung Disease (GOLD) (GOLD I-II).
3. BMI: obese class 1 (30-34.9).
4. Sex: male
5. They suffered from mild dyspnea, chronic cough and expectorations, with forced expiratory volume in one second (FEV1sec) from 50% to 80% of predicted value.

Exclusion criteria:

Patients with the following criteria will excluded from the study:

1. Severe psychiatric or cognitive impairments.
2. Progressive neuromuscular disorders.
3. Decreased level of consciousness.
4. Unstable fracture.
5. pacemaker inserted for fewer than 2 days
6. Deep-venous thrombosis (to minimize risk for pulmonary embolism from being in a prone position.
7. Mean arterial blood pressure of less than 65 mm Hg with or without vasopressors.
8. Tracheal surgery or sternotomy in the last 15 days.
9. Massive haemoptysis.
10. Intracranial pressure of more than 30 mm Hg or cerebral perfusion pressure of less than 60 mm Hg.

Ages: 50 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-02-17 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Pulmonary function test | One week for each comparator
  Spirometry is the most common pulmonary function test. It is widely used in the assessment of lung function to provide objective information used in the diagnosis of lung diseases and monitoring lung health Test started at the time of 20 minutes after subjects inhaling 400 μg of salbutamol. The following variables were assessed: FVC, FEV1, inspiratory capacity (IC), and inspiratory reserve volume (IRV)

CONTACTS AND LOCATIONS:
Overall Officials: Zahra Serry, Study Director — Faculty of physical therapy- internal medicine department
Locations (1):
- Cairo university- faculty of physical therapy, Cairo, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zakaria I, Serry ZMH, Soliman YMA, Aziz MM, Mohamed MI, Guirguis SA. Chest mobility exercises versus proprioceptive neuromuscular facilitation in patients with chronic obstructive pulmonary disease: A randomized trial. J Bodyw Mov Ther. 2025 Oct;44:400-408. doi: 10.1016/j.jbmt.2025.05.057. Epub 2025 Jun 4. PMID 40954608